CLINICAL TRIAL: NCT02874157
Title: Evaluation of Methods for Diagnosis of Cytomegalovirus Pneumonia in Mechanically Ventilated Patient
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-19; 2012-A00720-43 (Other: Ansm)
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: CMV Reactivation Diagnosis in ICU Patient
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: blood draw

SUMMARY:
Viral infections are only recently been investigated in patients on mechanical ventilation (MV) in ICU. It is especially the progress in the direct detection of these pathogens that allowed intensivists to try to assess objectively the impact of viruses in their patients. This is of course of viral infections "Community" (influenza virus, rhinovirus ...), but some viruses also occur under mechanical ventilation in immunocompetent adults. This is called viral infection "nosocomial" whose Herpesviridae are the most frequent and best studied. This replication Herpesviridae in ICU patients is usually a reactivation as primary infection. This reactivation is explained by the fact that after a few days of mechanical ventilation appears immunoparalysis, which can make the bed of bacterial or viral infection.Several studies have compared the pp65 antigenemia for quantitative PCR in immmunodéprimés patients. For example, in transplant patients (solid organs), the sensitivity of antigenemia was 91%, Quantitative PCR of 95.6% while the specificity was 57% and 81.6% respectively. No work, however, has to date compared these techniques in the intensive care patient. In a subject shortly epidemiological study, the sensitivity of the quantitative PCR performed on the LBA is 80%, when compared to antigenemia. Moreover this same study shows that half of the positive PCR on the BAL are not accompanied by a positive antigenemia, suggesting that PCR may be more sensitive than antigenemia. This exam has never been validated to date in intensive care. Finally, no work has so far evaluated the diagnostic performance of quantitative PCR performed on BAL

ELIGIBILITY:
Inclusion Criteria:

* Patient in ICU with ventilator-associated pneumonia suspicion

Exclusion Criteria:

* ICU pateint undergoing invasive ventilation for less than 48 hour

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patient undergoing invasive ventilation for more than 48h
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Number of CMV positive reactivation in ICU patient for sensitivity of quantitative PCR ( qPCR ) on LBA and CMV in whole blood compared with pp65 antigenemia. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille; Laurent PAPAZIAN, MD/PhD, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No